CLINICAL TRIAL: NCT01553851
Title: A Phase II Window of Opportunity Trial With GSK1120212 in Surgically Resectable Oral Cavity Squamous Cell Cancer
Brief Title: GSK1120212 in Surgically Resectable Oral Cavity Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201205124
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-10

CONDITIONS: Neoplasms, Oral; Mouth Neoplasms
MeSH Terms: conditions — Mouth Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1120212 (Experimental): GSK1120212 2 mg PO daily for a total of 14 days with the intent of the last pill being the day before surgery.
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — Trametinib (GSK1120212) is a selective MEK1 and MEK2 inhibitor with selective activity towards BRAF and RAS mutant cancer cell lines and hematopoietic cancer cells from AML and CML origins.
  Other Names: Trametinib; Mekinist

SUMMARY:
This phase II trial studies how trametinib effects tumor cells in patients with oral cavity squamous cell carcinoma that can be removed by surgery. Trametinib may shrink the tumor by blocking an enzyme pathway needed for cell growth.

DETAILED DESCRIPTION:
The rationale for this study in oral cavity squamous cell carcinomas rests on pre-clinical findings demonstrating that (a) activation of the ERK1/2 kinases is associated with aggressive features, (b) this aggressive phenotype is directly linked to expression of CD44, a cell surface hyaluronan receptor and (c) this association between activated ERK1/2 and CD44 is also identified in human cell lines and primary tumors. These data suggest that ERK1/2 is targetable biochemical pathway in CD44 expressing cells. These cells represent putative cancer stem cells or tumor initiating cells that have been associated with worse patient outcomes. Thus, the application of GSK1120212 to target OCSCC is a specific translational application of our laboratory findings.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed oral cavity squamous cell carcinoma of stage 2, 3, 4a, or 4b.
* Patients by definition have disease at the primary tumor site of at least 2 centimeters.
* Patient's treatment plan must include primary tumor site biopsy followed by gross excision of the primary tumor site at a separate operative procedure.
* Patients with concurrent primary head and neck tumors that will be resected as part of treatment plan are considered eligible
* Patients with head and neck cancer recurrence requiring surgery with no history of prior chemotherapy or radiation therapy are considered eligible.
* Patient must be ≥ 18 years of age.
* Patient must have an ECOG performance status ≤ 1
* Patient must have normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥1,200/mcl
  * Hemoglobin ≥9.0 g/dL
  * Platelets ≥100,000/mcl
  * PT/INR and PTT ≤1.3 x IULN (Subjects on Coumadin are included if their coagulation is within a normal therapeutic range)
  * LVEF ≥ILLN (by ECHO or MUGA)
  * Albumin ≥2.5 g/dL
  * Total bilirubin ≤1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 x IULN
  * Creatinine ≤1.5 x IULN OR Creatinine clearance ≥50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, intrauterine device, male partner sterilization, or complete abstinence) prior to study entry, for the duration of study participation, and for at least 4 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient must have the ability to swallow and retain orally administered medication.
* Patient (or legally authorized representative if applicable) must be able to understand and willing to sign an IRB approved written informed consent document.
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients must not have had any prior head and neck cancer treatment.
* Patient must not have a history of other malignancy ≤ 3 years previous with the exception of previous head and neck cancer treated only by surgery basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Patients must not be receiving any other investigational agents.
* Patient must not have a history of retinal vein occlusion (RVO).
* Patient must not have known symptomatic leptomeningeal or brain metastases or spinal cord compression.
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to GSK1120212 or other agents used in the study.
* Patient must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant and/or breastfeeding.
* Patient must not be known to be HIV-positive, hepatitis B-positive, or hepatitis C-positive (with the exception of chronic or cleared HBV or HCV infection, which will be allowed).
* Patient must not be taking any herbal supplements during the study (including but not limited to St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, or ginseng). If a potential patient is taking any herbal supplements, s/he must discontinue prior to beginning study treatment.
* Patient must not have any history or evidence of cardiovascular risk including any of the following:

  * QTcB ≥ 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: subjects with controlled atrial fibrillation for > 30 days prior to registration are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to registration
  * History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association.
  * Abnormal cardiac valve morphology (≥ grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
  * Treated refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic >90 mmHg which cannot be controlled by antihypertensive therapy.
  * Intra-cardiac defibrillator or permanent pacemaker
  * Cardiac metastases
* Patient must not have a history of interstitial lung disease or pneumonitis
* Current use of a prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Judd NP, Winkler AE, Murillo-Sauca O, Brotman JJ, Law JH, Lewis JS Jr, Dunn GP, Bui JD, Sunwoo JB, Uppaluri R. ERK1/2 regulation of CD44 modulates oral cancer aggressiveness. Cancer Res. 2012 Jan 1;72(1):365-74. doi: 10.1158/0008-5472.CAN-11-1831. Epub 2011 Nov 15. PMID 22086849
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK1120212
Started | 20
Completed | 17
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — constipation | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK1120212
Number analyzed (Participants) | 20
Age, Customized [Median (Full Range); unit: years]
  Median Age (years) | 59.5 [30 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
Oral Cavity Sub-Site [Number; unit: participants]
  Tongue | 7
  Floor of Mouth | 7
  Retromolar trigone | 5
  Buccal | 1
Clinical Stage [Number; unit: participants] — Cancer staging uses the TNM system where T=primary tumor, N stands for nodes (indicating cancer has spread to lymph nodes, and M for metastasis. Numbering associated with staging or letters denotes an increase in number, size, location or severity. Stage II (T2N0) Stage III (T2N1, T3N1) Stage IV(T2N2a,T2N2b,T3N2b,T4aN0,T4aN1,T4aN2b,T4aN2c)
  participants
    Stage II | 3
    Stage III | 3
    Stage IV | 14
History of Smoking and/or Alcohol Abuse [Number; unit: participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in Putative Tumor Initiating Cell Populations as Defined by Cell Surface CD44 and Intracellular Phospho-ERK1/2 Staining After Treatment With GSK1120212.
Description: Pre-post measure of p-EKP expression was measured by change in staining intensity and quartile distribution.
Time Frame: Baseline and Day 15
Population: Only15 of the 17 participants had sufficient pre- and post-treatment biopsies with sufficient tumor content to be evaluated for this biomarker assessment.
Measure: Number; unit: participants
Arm/Group | GSK1120212
Number analyzed (Participants) | 15
participants
  Decrease in p-EPK1/2 expression | 7
  Inverse relationship in p-EPK expression | 2
  No change in p-EKP expression | 3
  Increase in p-EKP expression | 3

2. Primary Outcome: Number of Participants With Changes in TumorCell Surface CD44 Expression After Treatment With GSK1120212.
Description: Pre-post measure of CD44 expression using IHC.
Time Frame: Baseline and Day 15
Measure: Number; unit: Participants
Arm/Group | GSK1120212
Number analyzed (Participants) | 15
Participants | 3

3. Secondary Outcome: Tumor Specific Findings for Pathologic Changes Including Proliferation (Ki-67 Staining), Tumor Vasculature Staining (Microvessel Density), ERK1/2 Mediated Changes in p27 (Kip1) & Flow Cytometric Analysis of the Peripheral Blood & Tumor.
Time Frame: Baseline and Day 15
Population: There was an insufficient amount of tissue to collected. The data was not collected and the outcome measure was not analyzed.
Arm/Group | GSK1120212
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Clinical Response Induced by GSK1120212, as Determined by Change in Tumor Size.
Description: Clinical Response was evaluted by quantitative changes in tumor size based on clinical examination of area of tumor at baseline and after GSK1120212 based on two dimensional measurements.
Time Frame: Baseline and Day 15
Measure: Number; unit: percentage of participants
Arm/Group | GSK1120212
Number analyzed (Participants) | 17
percentage of participants | 76

5. Secondary Outcome: Flow Cytometric Analysis of the Peripheral Blood and Tumor.
Description: Peripheral blood - baseline and Day 14
  Tumor - baseline and Day 15
Time Frame: Baseline, Day 14, and Day 15
Population: as for outcome 3
Arm/Group | GSK1120212
Number analyzed (Participants) | 0

6. Secondary Outcome: Percent Change in Maximum Standard Uptake Value in Oral Cavity Saqumous Cell Carcinoma (OCSCC) Using F18-Fluorodeoxyglucose-Positron Emission Tomography/Computed Tomography (FDG-PET/CT).
Time Frame: Baseline and Day 14
Population: Seven patients did not meet protocol-defined tumor size criteria (n=3), withdrew from study (n=3) or declined post GSK1120212 FDG-PET/CT(n=1)
Measure: Median (Full Range); unit: percentage change in SUVmax
Arm/Group | GSK1120212
Number analyzed (Participants) | 13
percentage change in SUVmax | -25 [-52 to -6]

7. Secondary Outcome: Safety of GSK1120212
Description: Number of adverse events were monitored for 30 day following last dose of GSK1120212
Time Frame: 1st 4-6 week follow-up visit
Measure: Number; unit: Adverse events
Arm/Group | GSK1120212
Number analyzed (Participants) | 20
Adverse events
  Neutrophil decrease (Grade 1-2) | 1
  Thrombocytopenia(Grade 1-2) | 1
  Colitis( Grade 3-4) | 1
  Diarrhea (Grade 1-2) | 3
  Mucositis( Grade 3-4) | 1
  Nausea (Grade 1-2) | 2
  Doudenal Perforation (Grade 3-4) | 1
  Stomach Cramps(Grade 1-2) | 1
  Lung Infection (Grade 3-4) | 1
  Rash, acneiform (Grade 1-2) | 9
  Pruritis (Grade 1-2) | 1
  Fatigue(Grade 1-2) | 2
  Fever (Grade 1-2) | 1
  Alkaline Phosphatase (Grade 1-2) | 3
  AST (Grade 1-2) | 4
  ALT (Grade 1-2) | 2
  Blurry Vision (Grade 1-2) | 1
  Hypotension (Grade 1-2) | 1

8. Secondary Outcome: Percent Change in Tumor Size Area
Time Frame: Baseline and Day 15
Population: Quantitative changes in tumor size based on clinical examination of area of tumor at baseline and after GSK1120212 based on two dimensional measurements.
Measure: Median (Full Range); unit: percent change in tumor size area
Arm/Group | GSK1120212
Number analyzed (Participants) | 17
percent change in tumor size area | -46 [-74 to -14]

9. Secondary Outcome: Percent of Participants With Metabolic Changes in OCSCC Using FDG-PET/CT Imaging.
Description: Intratumarol metabolic changes were evaluated by changes in in SUVmax in the primary tumor; quantitative analysis SUVmax with the primary tumor site was determined within a volume of interest around the tumor using a Siemens eSoft workstation.
Time Frame: Baseline and Day 14
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | GSK1120212
Number analyzed (Participants) | 13
percentage of participants | 85

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 4-6 weeks.
Description: AE grade 3 or higher will be followed for 3-6 months and considered at least possibly related
Arm/Group | GSK1120212
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 (N=20)
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood Bilirubin increased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White cell count decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 1
Duodenal Perforation (Gastrointestinal disorders) | 2
Sepsis (Infections and infestations) | 1
Infections and infestations -Other: Skin Infection (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 (N=20)
Anemia (Blood and lymphatic system disorders) | 9
Hypertension (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral Dysesthesia (Gastrointestinal disorders) | 1
Oral Hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 6
Small intestines obstruction (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Localized Edema (General disorders) | 1
Papulopustular rash (Infections and infestations) | 2
Infections and infestation-Other: Skin infection (Infections and infestations) | 1
Tracheostomy site bleed (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline Phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 1
Platelet count decreased (Investigations) | 5
Lymphocyte decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Small number of treated patients. Short duration of GSK1120212 administration. Biopsy limitations precluded analysis of all patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No